CLINICAL TRIAL: NCT06938854
Title: Prospective, Multi-center, Single-arm Investigational Study of SWM-831 to Treat Moderate and Severely Calcified Femoropopliteal Arteries
Brief Title: Investigational Study of SWM-831 to Treat Moderate and Severely Calcified Femoropopliteal Arteries
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Collaborators: Iqvia Pty Ltd (Industry); Massachusetts General Hospital (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 71411; jRCT2032240613 (Other: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: The objective of the study is to assess the safety and effectiveness of IVL to treat moderate and severely calcified femoropopliteal arteries, prior to DCB or stenting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Femoropopliteal Artery (Experimental): Up to 60 subjects with moderate or severely calcified femoropopliteal artery disease at up to 10 sites in Japan will be enrolled in the femoropopliteal clinical study. Destination therapy may include DCB or Stent based on post IVL assessment.
  In addition, a minimum of 10 and a maximum of 15 subjects with moderately or severely calcified iliac artery disease and a minimum of 10 and a maximum of 15 subjects with moderately or severely calcified BTK artery disease will also be enrolled to assess the safety and effectiveness of IVL in these two cohorts.
  Interventions: Device: Peripheral Intravascular Lithotripsy (IVL)

INTERVENTIONS:
Device: Peripheral Intravascular Lithotripsy (IVL) — For the Disrupt PAD Japan study, the Shockwave Medical Peripheral IVL System (SWM-831) is intended for lithotripsy enhanced balloon dilatation of lesions, including calcified lesions, in the peripheral vasculature, including the femoropopliteal arteries.
  Other Names: Intravascular Lithotripsy (IVL)

SUMMARY:
Disrupt PAD Japan is a prospective, multi-center, single-arm study of SWM-831 to treat moderate and severely calcified femoropopliteal arteries, prior to DCB or stenting.

DETAILED DESCRIPTION:
Up to 60 subjects at up to 10 sites in Japan will be enrolled in the femoropopliteal clinical study with moderate and severely calcified femoropopliteal artery disease presenting with Rutherford Category 2 - 5 of the target limb.

Two additional cohorts [Iliac and BTK (Below-the-Knee)] will enroll a minimum of 10 and a maximum of 15 subjects each with moderate and severely calcified iliac disease with a Rutherford Category (RC) 2 - 5 and a minimum of 10 and a maximum of 15 subjects with moderate and severely calcified BTK lesions with a Rutherford Category (RC) 2 - 5 will be enrolled and followed through 12 months.

The estimated study duration for these cohorts is approximately 24 months. Study subjects will be followed through discharge, 30 days, 6, and 12 months.

ELIGIBILITY:
General Inclusion Criteria:

Subjects are required to meet all of the following inclusion criteria in order to be enrolled in the clinical study:

1. Subject is able and willing to comply with all assessments in the study.
2. Subject or subject's legal representative has been informed of the nature of the study, agrees to participate and has signed the approved consent form.
3. Age of subject is ≥ 18. Note: If a subject is under 20 years, voluntary agreement shall be obtained from both the subject and the subject's representative or legal guardian using the written consent form.
4. Rutherford Clinical Category 2, 3, 4, or 5 of the target limb.
5. Estimated life expectancy > 1 year.

Angiographic Inclusion Criteria:

Subjects are required to meet all of the following inclusion criteria in order to be enrolled in the clinical study. For lesion characteristics, each target lesion must meet eligibility.

1. One target lesion that is located in a native, de novo superficial femoral artery (SFA) or popliteal artery (popliteal artery extends to and ends proximal to the ostium of the anterior tibial artery). <Not applicable to iliac or BTK cohort>
2. Target lesion reference vessel diameter (RVD) is between 4.0 mm and 8.0 mm by investigator visual estimate. <Not applicable to iliac or BTK cohort>
3. Target lesion with ≥ 70% stenosis by investigator visual estimate.
4. Target lesion length is ≤ 200 mm by investigator visual estimate. Target lesion can be all or part of the 200 mm treated zone.
5. Subject has at least one patent tibial vessel on the target limb with runoff to the foot, defined as no stenosis ≥ 50%.
6. Calcification is determined to be grade 2 - 4 (unilateral calcification ≥ 5 cm, bilateral wall calcification < 5 cm, and bilateral calcification ≥ 5 cm, respectively), as defined by PACSS (Peripheral Artery Calcification Scoring System). <Not applicable to iliac and BTK cohort>

Angiographic Inclusion Criteria specific to Iliac Arteries

1. Target lesion located in the native, de novo common or external iliac artery.
2. Target lesion reference vessel diameter (RVD) is between 5.0 mm and 10.0 mm by investigator visual estimate.
3. Evidence of PACSS calcification grade 2 - 4 and non-dilatable lesion indicating presence of calcium.

Note: Non-dilatable lesion requires attempted treatment with PTA during the index procedure with residual stenosis ≥ 50% and no serious angiographic complication.

Angiographic Inclusion Criteria specific to BTK Arteries

1. Target lesion from the native, de novo distal segment of the popliteal artery to the ankle joint.
2. Target lesion reference vessel diameter (RVD) is between 2.0 mm and 4.0 mm by investigator visual estimate.
3. Evidence of PACSS calcification grade 2 - 4 and non-dilatable lesion indicating presence of calcium.

Note: Non-dilatable lesion requires attempted treatment with PTA during the index procedure with residual stenosis ≥ 50% and no serious angiographic complication.

General Exclusion Criteria

Subjects who meet any of the following exclusion criteria may not be enrolled in the study:

1. Rutherford Clinical Category 0, 1 and 6.
2. Subject has known or suspected active infection evidenced by WBC > 14.0 (14000/mm3) within 14 days prior to index procedure.
3. Previous or planned target limb major amputation (above the ankle).
4. History of prior endovascular or surgical procedure on the index limb within the past 30 days or planned within 30 days of the index procedure.

   Note: Inflow treatment of non-target lesions is allowed provided successful treatment.
5. Subject in whom antiplatelet or anticoagulant therapy is contraindicated.
6. Subject has known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
7. Subject has known allergy to urethane, nylon, or silicone.
8. History of myocardial infarction within 60 days prior to enrollment.
9. History of stroke within 60 days prior to enrollment.
10. History of thrombolytic therapy within two weeks prior to enrollment.
11. Subject has acute or chronic renal disease with creatinine > 2.5 mg/dL, unless on dialysis.
12. Subject is pregnant or nursing.
13. Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint.
14. Subject has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.
15. The use of specialty balloons, re-entry or atherectomy devices.
16. Active COVID-19 or previously diagnosed COVID-19 with sequelae that could confound endpoint assessments.
17. Subject has an anticipated life span of less than one (1) year.

General Exclusion Criteria specific to BTK Arteries

1. Subjects with osteomyelitis or deep soft tissue infection in the target limb.
2. Acute limb ischemia (of either leg).
3. Occlusion of all the inframalleolar outflow arteries/vessels (i.e., desert foot) in the target limb.

Angiographic Exclusion Criteria

Subjects who meet any of the following exclusion criteria may not be enrolled in the study:

1. In-stent restenosis within 10 mm of the target lesion.
2. Lesion within 10 mm of the ostium of the SFA or within 10 mm proximal to the anterior tibial artery ostium. <Not applicable to iliac or BTK cohort>
3. Evidence of aneurysm or thrombus in target vessel.
4. No calcium or mild calcium in the target lesion by PACSS.
5. Target lesion within native or synthetic vessel grafts.
6. Subject has significant stenosis (≥ 50% stenosis) or occlusion of inflow tract before target treatment zone (e.g., iliac or common femoral) not successfully treated.
7. Failure to successfully treat significant distal non-target lesions, if treated prior to target lesion. Successful treatment is defined as obtaining < 50% residual stenosis with no serious angiographic complications (e.g., embolism).
8. Failure to successfully cross the guidewire across the target lesion; successful crossing defined as tip of the guidewire distal to the target lesion in the absence of flow limiting dissections or perforations.

Angiographic Exclusion Criteria specific to Iliac Arteries

1.Target lesion with any aorta involvement.

Angiographic Exclusion Criteria specific to BTK Arteries

1. Failure to treat clinically significant inflow lesions in the ipsilateral iliac, femoral, or popliteal arteries with < 30% residual stenosis, and no serious angiographic complications (e.g., embolism).
2. Treatment of vessels below the ankle joint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Subjects with Procedural Success | Day 0
  Primary Endpoint for Femoropopliteal: Procedural success is defined as residual stenosis < 50% without ≥ grade D dissections, prior to Drug-Coated Balloon (DCB) or stenting for the treated target lesion (core lab assessed)
Percentage of Subjects with Procedural Success | Day 0
  Primary Endpoint for Iliac: Procedural success is defined as residual stenosis < 50% without ≥ grade D dissections, prior to stenting for the treated target lesion (core lab assessed)
Percentage of Subjects with Procedural Success | Day 0
  Primary Endpoint for BTK: Procedural success is defined as final residual stenosis < 50% without ≥ grade D dissections for the treated target lesion (core lab assessed).

SECONDARY OUTCOMES:
Rate of ≥ grade D dissections, perforation, distal embolization, slow flow or acute vessel closure | Day 0
  Serious angiographic complications defined as the rate of ≥ grade D dissections, perforation, distal embolization, slow flow or acute vessel closure at the final procedural timepoint, as assessed by the angiographic core lab.
Residual stenosis < 50% without ≥ grade D dissections | Day 0
  Femoropopliteal Technical Success defined as residual stenosis < 50% without ≥ grade D dissections (core lab assessed) at the final timepoint (after DCB or stenting).
Residual stenosis < 30% without ≥ grade D dissections | Day 0
  Femoropopliteal Technical Success defined as residual stenosis < 30% without ≥ grade D dissections (core lab assessed) at the final timepoint (after DCB or stenting)
Number of participants with freedom from clinically-driven target lesion revascularization (CD-TLR) CEC adjudicated and freedom from restenosis as determined by duplex-derived peak systolic velocity ratio (PSVR) ≤ 2.4, assessed by the DUS core lab. | At 6 months and 12 months post-procedure
  Primary patency at 6 and 12 months defined as freedom from clinically-driven target lesion revascularization (CD-TLR) CEC adjudicated and freedom from restenosis as determined by duplex-derived peak systolic velocity ratio (PSVR) ≤ 2.4, assessed by the DUS core lab.
  - CD-TLR is defined as any revascularization (endovascular or surgical) within the target vessel due to symptoms or drop of ABI > 20% or > 0.15 when compared to the 30-day ABI and associated with an angiographic lesion ≥ 50% at the target lesion site.
Number of participants with Major Adverse Event | At 30 days, 6 months and 12 months post-procedure
  Major Adverse Event (MAE) at 30 days, 6 and 12 months Clinical Events Committee adjudicated (as a composite and individual components), defined as:
  - Cardiovascular death
  - Clinically-driven target lesion revascularization (CD-TLR)
  - Unplanned target limb major amputation (above the ankle)
Number of participants with change in Ankle brachial index (ABI) or Toe brachial index (TBI) | At 30 days, 6 months, and 12 months post-procedure
  Ankle brachial index (ABI) or Toe brachial index (TBI) at 30 days, 6, and 12 months reported as change from baseline
Number of participants with change in Rutherford Category | At 30 days, 6 months, and 12 months post-procedure
  Rutherford Category at 30 days, 6, 12 months reported as change from baseline

CONTACTS AND LOCATIONS:
Locations (10):
- Japan (10):
  - Asahi General Hospital, Asahi, Chiba
  - Tokyobay Urayasu Ichikawa, Chiba
  - Matsuyama Red Cross Hospital, Ehime
  - Kokura Memorial Hospital, Fukuoka
  - Caress Sapporo Tokeidai Memorial Hospital, Hokkaido
  - Tokushukai Shonan Kamakura General Hospital, Kanagawa
  - Sendai Kousei Hospital, Miyagi
  - Nara Medical University Hospital, Nara
  - Osaka International Medical & Science Center Daini Osaka Police Hospital, Osaka
  - Toho University Ohashi Medical Center, Tokyo

IPD SHARING:
Plan to Share IPD: No